CLINICAL TRIAL: NCT03229395
Title: Alterations of Muscle Secretome Associated With Muscle Atrophy Caused by Glucocorticoids
Acronym: MYOSECRET
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: UCL-MYOSECRET 2014-1
Record Dates: First submitted 2016-12-21; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2016-12

CONDITIONS: Cushing Syndrome
Keywords: skeletal muscle; muscle mass; glucocorticoids; biomarkers
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with Cushing's syndrome: Patients were selected by the PI at the diagnosis.
- control patients: Selected patients are matched for age and sex.

SUMMARY:
Several studies have shown that lean mass, in particular muscle mass, is an excellent predictive survival factor in many diseases. A better knowledge of the mechanisms responsible for muscle atrophy and the identification of atrophic process markers are deeply needed for the development of new anti-atrophic therapies. Either as drugs used to treat several medical conditions or as endocrine hormones released in response to many stress situations (e.g., sepsis, cancer, insulinopenia…), glucocorticoids (GC) are recognized to play a major role in skeletal muscle atrophy. Indeed, the inhibition of GC action by a receptor antagonist (RU486) or by muscle-specific invalidation of the GC receptor inhibits the muscle atrophy in these stress situations. Therefore, all these data clearly indicate that GC play a major role in skeletal muscle atrophy observed in several conditions. Emerging evidence has revealed that the skeletal muscle has a secretory function. Human skeletal muscle secretome was first estimated at about 300 proteins by computational analysis and proteomic analysis have recently confirmed these results. Some of these secreted proteins, conceptualized as myokines, can act locally on muscle cells through autocrine/paracrine loops and on surrounding tissues such as muscle blood vessels or can be released into the blood stream to produce systemic effects. One prominent example is interleukin (IL)-6 which is released into circulation by contracting skeletal muscle and can regulate metabolic and inflammatory processes. As IL-6, several other potential myokines have been identified including IL-8, IL-15, insulin-growth factor I (IGF-I), follistatin-like 1 (FSTL1) or fibroblast-growth factor (FGF)-21. Moreover, secreted proteins may also reflected metabolic changes which take place in muscle cells. Indeed, myoblast differentiation is accompanied by dramatic changes in the secreted proteins profile as increased expression of Semaphorins, IGF-I, matrix metalloproteinase (MMP)-2 or Collagens. Thereby, the investigators hypothesized that skeletal muscle atrophy induced by GC is associated with specific alterations of the muscle secretome. The aim of this project is to identify the GC-induced changes in the secretome of human skeletal muscle cells in culture (in vitro approach) and to determine how these changes translate into the circulation of subjects exposed to high concentrations of GC (Cushing's syndrome) (in vivo approach). Characterization of these changes in human subjects should allow to better understand the cellular mechanisms involved in muscle atrophy and might lead to identify circulating biomarkers associated with skeletal muscle atrophy, as telopeptides are for bone tissue.

ELIGIBILITY:
Inclusion Criteria:

* Pituitary or adrenal endogenous Cushing's syndrome formally demonstrated by the standard endocrinological assessment
* New diagnosis or recurrence or persistent Cushing's syndrome after pituitary surgery

Exclusion Criteria:

* Pseudo Cushing's syndrome
* Paraneoplasic Cushing's syndrome
* Cyclic Cushing's syndrome
* Adrenocortical carcinoma
* Pituitary irradiation during the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Cushing's syndrome are caracterised by elevated circulating glucocorticoid levels generally due to a pitiutary or adrenal adenoma. These patients were compared to heathly control patients who are matched for age and sex.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Measurement of BMI in kg/m^2 | 1 day (one assessment at diagnosis)
  Measurement of weight in kilograms and height in meters to determine BMI as BMI=weight/height^2
Evaluation of quality of life of Cushing's patients | 1 day (one assessment at diagnosis)
  The CushingQoL questionnaire was used to evaluate quality of life of Cushing's patients
Measure of body lean mass of Cushing's and control patients | 1 day (one assessment at diagnosis)
  Bioelectrical Impedance Vector Analysis (BIA) was used for evaluation of lean and fat mass.
Muscle strenght measurement of Cushing's and control patients | 1 day (one assessment at diagnosis)
  Evalutation by dynamometer "Jamar type"
Measurement of Mid-arm muscle circumference (MAMC, cm) | 1 day (one assessment at diagnosis)
  Measurement of triceps skinfold thickness (TSF, in cm), and midarm circumference (MAC, in cm) to determine the MAMC according to the following formula: MAMC= MAC - (Pi x TSF).
  MAMC is a bedside anthropometric measurement that estimates somatic protein reserve, an early indicator of nutritional depletion.
Evaluation of daily energy expenditure (DEE) of Cushing's and control patients | 1 day (one assessment at diagnosis)
  Evaluation of DEE by completing the QAPSE questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marie De Barsy, Nurse, Study Chair — Cliniques Universitaires St Luc
Locations (1):
- De Barsy Marie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen BK. Muscle as a secretory organ. Compr Physiol. 2013 Jul;3(3):1337-62. doi: 10.1002/cphy.c120033. PMID 23897689
- [Background] Schakman O, Kalista S, Barbe C, Loumaye A, Thissen JP. Glucocorticoid-induced skeletal muscle atrophy. Int J Biochem Cell Biol. 2013 Oct;45(10):2163-72. doi: 10.1016/j.biocel.2013.05.036. Epub 2013 Jun 24. PMID 23806868
- [Background] Stastna M, Van Eyk JE. Secreted proteins as a fundamental source for biomarker discovery. Proteomics. 2012 Feb;12(4-5):722-35. doi: 10.1002/pmic.201100346. Epub 2012 Jan 19. PMID 22247067
- [Result] Baracos VE, Reiman T, Mourtzakis M, Gioulbasanis I, Antoun S. Body composition in patients with non-small cell lung cancer: a contemporary view of cancer cachexia with the use of computed tomography image analysis. Am J Clin Nutr. 2010 Apr;91(4):1133S-1137S. doi: 10.3945/ajcn.2010.28608C. Epub 2010 Feb 17. PMID 20164322
- [Result] Bortoluzzi S, Scannapieco P, Cestaro A, Danieli GA, Schiaffino S. Computational reconstruction of the human skeletal muscle secretome. Proteins. 2006 Mar 15;62(3):776-92. doi: 10.1002/prot.20803. PMID 16342272
- [Result] Braun TP, Grossberg AJ, Krasnow SM, Levasseur PR, Szumowski M, Zhu XX, Maxson JE, Knoll JG, Barnes AP, Marks DL. Cancer- and endotoxin-induced cachexia require intact glucocorticoid signaling in skeletal muscle. FASEB J. 2013 Sep;27(9):3572-82. doi: 10.1096/fj.13-230375. Epub 2013 Jun 3. PMID 23733748
- [Result] Gueugneau M, Coudy-Gandilhon C, Theron L, Meunier B, Barboiron C, Combaret L, Taillandier D, Polge C, Attaix D, Picard B, Verney J, Roche F, Feasson L, Barthelemy JC, Bechet D. Skeletal muscle lipid content and oxidative activity in relation to muscle fiber type in aging and metabolic syndrome. J Gerontol A Biol Sci Med Sci. 2015 May;70(5):566-76. doi: 10.1093/gerona/glu086. Epub 2014 Jun 17. PMID 24939997
- [Result] Henningsen J, Rigbolt KT, Blagoev B, Pedersen BK, Kratchmarova I. Dynamics of the skeletal muscle secretome during myoblast differentiation. Mol Cell Proteomics. 2010 Nov;9(11):2482-96. doi: 10.1074/mcp.M110.002113. Epub 2010 Jul 14. PMID 20631206
- [Result] Hu Z, Wang H, Lee IH, Du J, Mitch WE. Endogenous glucocorticoids and impaired insulin signaling are both required to stimulate muscle wasting under pathophysiological conditions in mice. J Clin Invest. 2009 Oct;119(10):3059-69. doi: 10.1172/JCI38770. Epub 2009 Sep 14. PMID 19759515
- [Result] Le Bihan MC, Bigot A, Jensen SS, Dennis JL, Rogowska-Wrzesinska A, Laine J, Gache V, Furling D, Jensen ON, Voit T, Mouly V, Coulton GR, Butler-Browne G. In-depth analysis of the secretome identifies three major independent secretory pathways in differentiating human myoblasts. J Proteomics. 2012 Dec 21;77:344-56. doi: 10.1016/j.jprot.2012.09.008. Epub 2012 Sep 20. PMID 23000592
- [Result] Mourtzakis M, Prado CM, Lieffers JR, Reiman T, McCargar LJ, Baracos VE. A practical and precise approach to quantification of body composition in cancer patients using computed tomography images acquired during routine care. Appl Physiol Nutr Metab. 2008 Oct;33(5):997-1006. doi: 10.1139/H08-075. PMID 18923576
- [Result] Neves M Jr, Barreto G, Boobis L, Harris R, Roschel H, Tricoli V, Ugrinowitsch C, Negrao C, Gualano B. Incidence of adverse events associated with percutaneous muscular biopsy among healthy and diseased subjects. Scand J Med Sci Sports. 2012 Apr;22(2):175-8. doi: 10.1111/j.1600-0838.2010.01264.x. Epub 2011 Mar 10. PMID 21392121
- [Result] Piccoli A. Patterns of bioelectrical impedance vector analysis: learning from electrocardiography and forgetting electric circuit models. Nutrition. 2002 Jun;18(6):520-1. doi: 10.1016/s0899-9007(02)00771-2. No abstract available. PMID 12044826
- [Result] Schakman O, Dehoux M, Bouchuari S, Delaere S, Lause P, Decroly N, Shoelson SE, Thissen JP. Role of IGF-I and the TNFalpha/NF-kappaB pathway in the induction of muscle atrogenes by acute inflammation. Am J Physiol Endocrinol Metab. 2012 Sep 15;303(6):E729-39. doi: 10.1152/ajpendo.00060.2012. Epub 2012 Jun 26. PMID 22739109
- [Result] Webb SM, Badia X, Barahona MJ, Colao A, Strasburger CJ, Tabarin A, van Aken MO, Pivonello R, Stalla G, Lamberts SW, Glusman JE. Evaluation of health-related quality of life in patients with Cushing's syndrome with a new questionnaire. Eur J Endocrinol. 2008 May;158(5):623-30. doi: 10.1530/EJE-07-0762. PMID 18426820